CLINICAL TRIAL: NCT02007044
Title: Ibrutinib vs Ibrutinib + Rituximab (i vs iR) in Patients With Relapsed (CLL)
Brief Title: Ibrutinib With or Without Rituximab in Treating Patients With Relapsed Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0703; NCI-2014-00989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2014-00843; 2013-0703 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (ibrutinib, rituximab) (Experimental): Patients receive ibrutinib as in Arm I beginning on day 1 or 2. Patients also receive rituximab IV over 3-8 hours on days 1, 8, 15, and 22 of cycle 1 and day 1 of cycles 2-6. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
  Arms: Arm II (ibrutinib, rituximab)

SUMMARY:
This phase II trial studies ibrutinib with or without rituximab in treating patients with chronic lymphocytic leukemia that has come back after treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether ibrutinib is more effective with or without rituximab in treating chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 2-year progression-free survival (PFS) rate in treated patients.

SECONDARY OBJECTIVE:

I. To determine safety and tolerability, the overall response rate (ORR), the estimated PFS, changes in immune parameters (lymphocyte subpopulations, immunoglobulin levels) and biomarker responses in relapsed chronic lymphocytic leukemia (CLL) patients receiving ibrutinib (i) versus ibrutinib and rituximab (iR).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ibrutinib as in Arm I beginning on day 1 or 2. Patients also receive rituximab intravenously (IV) over 3-8 hours on days 1, 8, 15, and 22 of cycle 1 and day 1 of cycles 2-6. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 60 days and then every 4 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of CLL/small lymphocytic lymphoma (SLL) or prolymphocytic leukemia (PLL) and be previously treated; given the poor outcome of CLL/SLL/PLL patients with 17p deletion (del) or tumor protein (TP)53 mutation to standard frontline chemo-immunotherapy, such patients will be eligible if they are untreated
* Patients must have an indication for treatment by 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria
* Patients must be age >= 18 years at the time of signing informed consent, understand and voluntarily sign an informed consent, and be able to comply with study procedures and follow-up examinations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients of childbearing potential must be willing to practice highly effective birth control (e.g., condoms, implants, injectables, combined oral contraceptives, intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the study and for 30 days after the last dose of study drug; women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) except for patients with bilirubin elevation due to Gilbert's disease who will be allowed to participate
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft-Gault equation unless disease related
* Free of prior malignancies for 3 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast, who are eligible even if they are currently treated or have been treated and/or diagnosed in the past 3 years prior to study enrollment; if patients have another malignancy that was treated within the last 3 years, such patients can be enrolled, after consultation with the principal investigator, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center
* A urine pregnancy test (within 7 days of enrollment date) is required for women with childbearing potential

Exclusion Criteria:

* Pregnant or breast-feeding females
* Prior therapy with ibrutinib or other kinase inhibitors that target Bruton's tyrosine kinase (BTK); patients who previously received therapy with the phosphoinositide-3 kinase (PI3K) delta inhibitor idelalisib (Zydelig) are allowed to be enrolled
* Treatment including chemotherapy, chemo-immunotherapy, monoclonal antibody therapy, radiotherapy, high-dose corticosteroid therapy (more than 60 mg prednisone daily or equivalent), or immunotherapy within 21 days prior to enrollment or concurrent with this trial
* Investigational agent received within 30 days prior to the first dose of study drug
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Patients with uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP)
* Patients with severe hematopoietic insufficiency, as defined by an absolute neutrophil count of less than 500/uL, unless disease-related, and/or a platelet count of less than 30,000/uL at time of screening for this protocol
* Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo therapy with ibrutinib and rituximab
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* History of stroke or cerebral hemorrhage within 6 months
* Evidence of bleeding diathesis or coagulopathy within 3 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment date, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to enrollment date; bone marrow aspiration and/or biopsy are allowed
* Serious, non-healing wound, ulcer, or bone fracture
* Treatment with Coumadin; patients who recently received Coumadin must be off Coumadin for at least 7 days prior to start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-12-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | Time from start of treatment to progression or death date, assessed at 2 years
  A two-sided log-rank test will be used to assess the differences of progression-free survival between the treatment groups.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Toxicity will be reported by type, frequency and severity. Highest toxicity grades per patient per course will be tabulated for selected adverse events and laboratory measurements.
Overall response rate | Up to 5 years
  Wilcoxon rank test will be used in the data analyses of continuous variables.
Estimated progression-free survival | Up to 5 years
  Time to progression functions will be estimated using the Kaplan-Meier method. A two-sided log-rank test will be used to assess the differences of progression-free survival between the treatment groups.
Changes in immune parameters (lymphocyte subpopulations, immunoglobulin levels) | Baseline to up to 5 years
  Will be assessed by flow cytometry.
Quality of life (QOL) | Up to 24 cycles (96 weeks)
  Will be assessed by the European Organization for Research and Treatment of Cancer QOL Questionnaire (EORTC QLQ-C30). Analyzed by linear mixed models for longitudinal data. These models allow each patient to have a random intercept and a random slope, which describe their differences at baseline and their different changing trends over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Burger, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Burger JA, Sivina M, Jain N, Kim E, Kadia T, Estrov Z, Nogueras-Gonzalez GM, Huang X, Jorgensen J, Li J, Cheng M, Clow F, Ohanian M, Andreeff M, Mathew T, Thompson P, Kantarjian H, O'Brien S, Wierda WG, Ferrajoli A, Keating MJ. Randomized trial of ibrutinib vs ibrutinib plus rituximab in patients with chronic lymphocytic leukemia. Blood. 2019 Mar 7;133(10):1011-1019. doi: 10.1182/blood-2018-10-879429. Epub 2018 Dec 7. PMID 30530801
- See also: MD Anderson Cancer Center — http://www.mdanderson.org